CLINICAL TRIAL: NCT03562897
Title: Efficacy of the Oncoxin-Viusid® Nutritional Supplement on the Quality of Life of Patients With Advanced or Metastatic Ovarian Epithelial Cancer. Clinical Trial Phase II.
Brief Title: Evaluation of Ocoxin-Viusid® in Advanced or Metastatic Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-7
Record Dates: First submitted 2018-05-25; First posted 2018-06-20 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-10

CONDITIONS: Carcinoma; Ovarian Neoplasm; Endocrine Gland Neoplasm; Urogenital Neoplasms; Ovarian Diseases; Adnexal Diseases; Genital Diseases, Female; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Endocrine System Diseases; Gonadal Disorders; Genital Neoplasm, Female; Neoplasms, Glandular and Epithelial
Keywords: Dietary supplements; Ocoxin-Viusid; Nutritional supplement; Ovarian Cancer; Metastasis
MeSH Terms: conditions — Carcinoma; Ovarian Neoplasms; Endocrine Gland Neoplasms; Urogenital Neoplasms; Ovarian Diseases; Adnexal Diseases; Genital Diseases, Female; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Endocrine System Diseases; Gonadal Disorders; Genital Neoplasms, Female; Neoplasms, Glandular and Epithelial; Neoplasm Metastasis | interventions — Ocoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocoxin-Viusid® (Experimental): Ocoxin-Viusid® before, during and after the Chemotherapy treatment.
  Interventions: Dietary Supplement: Ocoxin-Viusid

INTERVENTIONS:
Dietary Supplement: Ocoxin-Viusid — Ocoxin-Viusid group (Experimental): Oral solution Ocoxin-Viusid (30 ml vials) were used at a rate of 60ml / day (1 vial every 12 hours), preferably administered after breakfast and dinner. The treatment will start a week before start Chemotheray treatment (CT) and, It will maintenance until 3 weeks after finished the last cycle of CT (3 cycles of CT of Carboplatin/Paclitaxel or Cisplatin/ Paclitaxel with neoadjuvant intent).

SUMMARY:
Our hypothesis is: the nutritional supplement Ocoxin-viusid improves the quality of life of patients, including a better tolerance to neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
General Objectives -To identify the efficacy of the nutritional supplement Ocoxin-viusid to increase the quality of life of patients with epithelial advanced or metastatic ovarian cancer. Specific Objectives - Identify the influence of the research product on the nutritional status and quality of life of patients. - Describe the toxicity of the research product. - Identify the adverse reactions to the chemotherapy scheme and quantify the interruptions to it by acute toxicity.

Quality of life. It will be measured as: - EORTC Questionnaire QLQ-C30 (Score of each item and general score). Measurement time: at the beginning and 3 weeks after the 3rd cycle of QT - EORTC Questionnaire QLQ-OV28 (Score of each item and general score). Measurement time: at the beginning and 3 weeks after the 3rd cycle of QT - Karnofsky index (Score of 0-100 points at intervals of 10). Measurement time: at the beginning, in each cycle of QT and 3 weeks after the 3rd cycle of QT

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 years of age or older.
2. Patients with diagnosis of ovarian epithelial cancer in stages III (not resectable) and IV.
3. Patients with general health status according to the Karnofsky Index ≥ 70 (Annex 12).
4. Life expectancy equal to or greater than 3 months.
5. Patients who give their informed consent in writing to participate in the study.
6. Normal functioning of organs and bone marrow defined by the following parameters: -Hemoglobin ≥ 90 g / L - Total Leukocyte count ≥ 3.0 x 109 / L Absolute Neutrophil Count = 1.5 x 109 / L -Platelet count ≥ 100 x 109 / L -Glycemia values ≤ 10 Umol / L -Values of Creatinine and total bilirubin within the normal limits of the institution. -Values of AST / ALT ≤2.5 times the upper limit of the normal interval established in the institution.
7. Patients with a history of cardiovascular disease, with ejection fraction ≥ 55%, measured by echocardiogram.

Exclusion Criteria:

1. Patients who are receiving another research product.
2. Patients with known hypersensitivity to QT with Carboplatin, Cisplatin and / or Paclitaxel.
3. Patients in stage III tributary of surgical treatment at diagnosis.
4. Patients with known hypersensitivity to any ingredient of the product research.
5. Decompensated intercurrent diseases, including: active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, liver diseases and psychiatric illnesses that could limit adherence to the requirements of the clinical trial or any other special condition that at the discretion of the physician put your health or life at risk during your participation in the trial.
6. Pregnancy, breastfeeding or puerperium.
7. Patients with brain metastases and/or leptomeningeal carcinosis.
8. Patients' carrier of the human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 months
  It will measured by: - EORTC QLQ-C30 (Points of every item and final points)
Quality of life | 4 months
  Karnofsky index (Score of 0-100 points at intervals of 10)
Quality of life | 4 months
  EORTC QLQ-OV28 (Points of every item and final points)

SECONDARY OUTCOMES:
Nutritional State | 4 months
  Body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology and Radiobiology (INOR), Havana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Prat J. New insights into ovarian cancer pathology. Ann Oncol. 2012 Sep;23 Suppl 10:x111-7. doi: 10.1093/annonc/mds300. PMID 22987944
- [Background] Jelovac D, Armstrong DK. Recent progress in the diagnosis and treatment of ovarian cancer. CA Cancer J Clin. 2011 May-Jun;61(3):183-203. doi: 10.3322/caac.20113. Epub 2011 Apr 26. PMID 21521830
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Landen CN Jr, Birrer MJ, Sood AK. Early events in the pathogenesis of epithelial ovarian cancer. J Clin Oncol. 2008 Feb 20;26(6):995-1005. doi: 10.1200/JCO.2006.07.9970. Epub 2008 Jan 14. PMID 18195328
- [Background] Fuchs-Tarlovsky V, Alvarez-Altamirano K, Turquie-Sacal D, Alvarez-Flores C, Hernandez-Steller H. Nutritional status and body composition are already affected before oncology treatment in ovarian cancer. Asia Pac J Clin Nutr. 2013;22(3):426-30. doi: 10.6133/apjcn.2013.22.3.12. PMID 23945413
- [Background] Gupta D, Lis CG, Vashi PG, Lammersfeld CA. Impact of improved nutritional status on survival in ovarian cancer. Support Care Cancer. 2010 Mar;18(3):373-81. doi: 10.1007/s00520-009-0670-y. Epub 2009 May 31. PMID 19484479
- [Background] Kathiresan AS, Brookfield KF, Schuman SI, Lucci JA 3rd. Malnutrition as a predictor of poor postoperative outcomes in gynecologic cancer patients. Arch Gynecol Obstet. 2011 Aug;284(2):445-51. doi: 10.1007/s00404-010-1659-y. Epub 2010 Aug 29. PMID 20803205
- [Background] Madhok BM, Yeluri S, Haigh K, Burton A, Broadhead T, Jayne DG. Parenteral nutrition for patients with advanced ovarian malignancy. J Hum Nutr Diet. 2011 Apr;24(2):187-91. doi: 10.1111/j.1365-277X.2010.01127.x. PMID 21843153
- [Background] Billson HA, Holland C, Curwell J, Davey VL, Kinsey L, Lawton LJ, Whitworth AJ, Burden S. Perioperative nutrition interventions for women with ovarian cancer. Cochrane Database Syst Rev. 2013 Sep 11;2013(9):CD009884. doi: 10.1002/14651858.CD009884.pub2. PMID 24027084
- [Background] Lohsiriwat V. The influence of preoperative nutritional status on the outcomes of an enhanced recovery after surgery (ERAS) programme for colorectal cancer surgery. Tech Coloproctol. 2014 Nov;18(11):1075-80. doi: 10.1007/s10151-014-1210-4. Epub 2014 Sep 13. PMID 25216721
- [Background] Andreyev HJ, Norman AR, Oates J, Cunningham D. Why do patients with weight loss have a worse outcome when undergoing chemotherapy for gastrointestinal malignancies? Eur J Cancer. 1998 Mar;34(4):503-9. doi: 10.1016/s0959-8049(97)10090-9. PMID 9713300
- [Background] Lamson DW, Brignall MS. Antioxidants in cancer therapy; their actions and interactions with oncologic therapies. Altern Med Rev. 1999 Oct;4(5):304-29. PMID 10559547
- [Background] Lamson DW, Brignall MS. Natural agents in the prevention of cancer, part two: preclinical data and chemoprevention for common cancers. Altern Med Rev. 2001 Apr;6(2):167-87. PMID 11302780
- [Background] Al-Mahtab M, Akbar SM, Khan MS, Rahman S. Increased survival of patients with end-stage hepatocellular carcinoma due to intake of ONCOXIN(R), a dietary supplement. Indian J Cancer. 2015 Jul-Sep;52(3):443-6. doi: 10.4103/0019-509X.176699. PMID 26905163